CLINICAL TRIAL: NCT00016328
Title: A Phase II Study of CCI-779 in Patients With Recurrent Glioblastoma Multiforme
Brief Title: CCI-779 in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01858; N997B; CDR0000068623; NCCTG-N997B; U10CA025224 (NIH)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-06

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive CCI-779 IV over 30 minutes once weekly for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
Phase II trial to study the effectiveness of CCI-779 in treating patients who have recurrent glioblastoma multiforme. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of CCI-779, in terms of the percentage of patients who are progression-free at 6 months, time to progression, and time to death, in patients with recurrent glioblastoma multiforme.

II. Determine the toxic effects of this drug in these patients. III. Correlate molecular alterations in the tumors of these patients with response to treatment with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to concurrent P450 anticonvulsant use (yes vs no).

Patients receive CCI-779 IV over 30 minutes once weekly for 4 weeks. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 6 months for 5 years and then annually for up to 10 years.

PROJECTED ACCRUAL: A total of 63 patients will be accrued for this study within 39 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed grade 4 astrocytoma at primary diagnosis or recurrence

  * Gliosarcoma allowed
* Evidence of tumor progression by MRI or CT scan after radiotherapy or first-line chemotherapy
* Measurable or evaluable disease by MRI or CT scan
* Performance status - ECOG 0-2
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL
* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3 times upper limit of normal
* Creatinine no greater than 2.0 mg/dL
* No myocardial infarction within the past 6 months
* No congestive heart failure requiring ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Cholesterol no greater than 350 mg/dL
* Triglycerides no greater than 400 mg/dL
* Willing to provide correlative laboratory samples
* No uncontrolled infection
* No known hypersensitivity to any components of CCI-779, diphenhydramine hydrochloride, or other similar antihistamines
* No other medical reason that would preclude diphenhydramine premedication
* No other active malignancy
* No other severe disease that would preclude study participation
* Not immunocompromised unless due to corticosteroids
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* See Disease Characteristics
* Prior adjuvant chemotherapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No more than 1 prior chemotherapy regimen for recurrent/progressive disease
* No prior polifeprosan 20 with carmustine implant (Gliadel)
* Must be on fixed dose of corticosteroids (or no corticosteroids) at least 1 week prior to baseline scan
* See Disease Characteristics
* At least 12 weeks since prior radiotherapy
* No prior stereotactic radiosurgery or interstitial brachytherapy unless there is a separate lesion on MRI that is outside of the previously treated field
* No prior resection since last chemotherapy or radiotherapy unless there is unequivocal tumor growth on neuro-imaging study since surgery or there is a separate lesion not present in the surgical bed
* More than 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2001-05; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients being progression free | 6 months
  Ninety-five percent confidence intervals for the true proportion will be calculated according to the approach of Duffy and Santner.

SECONDARY OUTCOMES:
Percentage of patients that have not progressed | 3 months
  Ninety-five percent confidence intervals for the true proportion will be calculated according to the approach of Duffy and Santner.
Percentage of patients that have not progressed | 12 months
  Ninety-five percent confidence intervals for the true proportion will be calculated according to the approach of Duffy and Santner.
Percentage of patients that have not progressed | 18 months
  Ninety-five percent confidence intervals for the true proportion will be calculated according to the approach of Duffy and Santner.
Confirmed tumor response defined as an objective status of complete response (CR), partial response (PR), or regression (REGR) on two consecutive evaluations | Up to 10 years
  Ninety-five percent confidence intervals for the true proportion will be calculated using the exact binomial method.
Time to progression and death | Up to 10 years
  Estimated using Kaplan-Meier. Frequency distributions of baseline patient characteristics will be compared using chi-squared and Wilcoxon tests.

CONTACTS AND LOCATIONS:
Overall Officials: Evanthia Galanis, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States